CLINICAL TRIAL: NCT05084885
Title: The Context of Gambling Treatment: Towards Creating an Online Service to Reduce Problem Gambling - Part Five
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 074-2018
Record Dates: First submitted 2019-08-14; First posted 2021-10-20 (Actual); Results first posted 2022-08-01 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Problem Gambling

STUDY DESIGN:
Intervention Model Description: The study will be evaluated using a pre-test vs. post-test design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online treatment (Experimental): The participants will receive counseling over the internet.
  Interventions: Other: Online therapy
- Non-treatment (No Intervention): Participants who did not participant in the group were asked to complete the 12ve month followup questionnaire (but not the post treatment questionnaire).

INTERVENTIONS:
Other: Online therapy — Standard counseling provided over the internet.
  Arms: Online treatment

SUMMARY:
This application involves a multi-stage study with the ultimate goal of developing an online treatment service for problem gamblers. We will recruit up to 100 problem gamblers, and offer problem gambling treatment services to them entirely over the internet. The program will be evaluated based on uptake, experience of the participants, and pre-test vs post-test differences in gambling and well-being.

DETAILED DESCRIPTION:
Disordered gambling is now recognized as a behavioral addiction. Although the physical consequences of the disorder are very mild, the financial and emotional costs can be enormous. This application involves a multi-stage study with the ultimate goal of developing an online treatment service for problem gamblers. This project was originally designed to take place over a three-year period but has been condensed into two. Part one was scoping review. Part two involved focus groups with service providers and people experiencing gambling problems. Part three will gather some general population information on two on going population survey's run by our research team. Part four Involved key informant interviews, and part five would be the development and evaluation of a pilot online treatment service. This application deals with part five of the overall project, Parts two and four were conducted as 025-2017. In this study, we will recruit up to 100 problem gamblers, and offer problem gambling treatment services to them entirely over the internet. The program will be evaluated based on uptake, experience of the participants, and pre-test vs post-test differences in gambling and well-being. The data reported here are related to part 5 only. Due to funding cuts, we were only able to include 2 people in the completed study.

ELIGIBILITY:
Inclusion Criteria:

* problem gamblers seeking treatment who are 18 years and older must be willing to have therapy conducted online must have access to a computer and Internet be able to communicate in English.

Exclusion Criteria:

* not able to communicate in English, has current suicidal ideation, acute psychotic symptoms, current involvement in other gambling treatment, has severe substance abuse problem or complex mental health problems (as assessed by screening tools)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2020-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nigel E Turner, Ph.D, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared with other researchers.

RESULTS

PARTICIPANT FLOW:
Groups:
- Non Treatment: Receive no treatment
Period: Baseline
Arm/Group | Online Treatment | Non Treatment
Started | 3 | 13
Treated | 2 | 0
Not Treated | 1 | 13
Completed | 2 | 13
Not Completed | 1 | 0
Period: Post Treatment
Arm/Group | Online Treatment | Non Treatment
Started | 2 | 13
Completed | 2 | 13
Not Completed | 0 | 0
Period: Follow-up
Arm/Group | Online Treatment | Non Treatment
Started | 2 | 13
Treated | 2 | 0
Not Treated | 0 | 13
Completed | 2 | 8
Not Completed | 0 | 5

BASELINE CHARACTERISTICS:
Arm/Group | Online Treatment
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Changes in Gambling Frequency as Measured by Self Reported Frequency on 12 Different Types of Gambling.
Description: Level of gambling frequency was measured using self reported frequency on a 7 point scale on 12 types of gambling. We used the maximum frequency across the twelve types of gambling so that if they reported participating in 5 types of gambling ranging from once per year (score of 1) to everyday (score of 7), we would score the person as 7. This way the measure was sensitive to changes in the most problematic frequent form of gambling for that person. Lower levels of gambling frequency after 12 months would be a positive outcome. To score frequency we computed each person's highest frequency for a range from 0 (none) to 7 (everyday) with higher numbers indicating more frequent gambling. The same was done for their post-test scores. We computed the difference score of post-test from pre-test which could range from 7 to -7 with negative numbers indicating improvement (reduced gambling participation).
Time Frame: Change from baseline to 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Treatment
Number analyzed (Participants) | 2
score on a scale | -2 (1.41)

2. Primary Outcome: Changes in Problem Gambling Severity Index (PGSI; Ferris & Wynne, 2001).
Description: Gambling problems are measured using PGSI (Ferris & Wynne, 2001). Each of the 9 item is measured on a 4 point scale from never (0) to almost always (3). The total ranges from 0 to 27. Higher scores indicate more gambling problems; Lower scores at followup would be a positive outcome. Total scores form 3 to 7 indicate moderate gambling problems; scores 7 or higher indicate severe gambling problems. In this study we subtracted pre-test scores from post test scores to compute a change score which would range from27 to -27 with higher number indicating a worse outcome and negative numbers indicating a positive outcome.
Time Frame: Change from baseline to 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Treatment
Number analyzed (Participants) | 2
score on a scale | -6 (1.41)

3. Primary Outcome: Changes in Kessler-6 (K6; Galea, et al., 2007).
Description: The Kessler-6 measures psychological distress (K6; Galea, et al., 2007). Higher scores indicate more psychological distress. Score 0 to 25 with scores over 8 indicating moderate psychological distress. We are predicting lower levels of psychological distress at 3 follow-up as measured using the Kessler-6 (K6; Galea, et al., 2007). For the evaluation we computed the difference of post-test from pre-test with a range from 25 to -25 with negative numbers indicating an improvement.
Time Frame: Change from baseline to 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Online Treatment
Number analyzed (Participants) | 2
units on a scale | -2 (0)

4. Primary Outcome: Changes in Mindful Attention Awareness Scale (MAAS; Brown & Ryan, 2003).
Description: Mindfulness was measured using the Mindful Attention Awareness Scale (MAAS; Brown & Ryan, 2003). Range 1 to 6 based on average score per item; higher scores mean greater mindfulness. For the evaluation we computed the difference of the post-test and the pre-test for a range from 6 to -6 with positive numbers indicating an improvement in mindfulness.
Time Frame: Change from baseline to 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Treatment
Number analyzed (Participants) | 2
score on a scale | .6 (.19)

5. Primary Outcome: Changes in Number of Games Played
Description: Number of games played was measured using a self report measure of participation in 12 games (see frequently above). Fewer games played would be a positive outcome. Possible range is from 0 to 12. We computed the difference score from pre-test to post-test which could range from 12 to -12 with negative numbers indicating improvement (reduced gambling participation).
Time Frame: Change from baseline to 3 months
Measure: Mean (Standard Deviation); unit: changes in number of games played
Arm/Group | Online Treatment
Number analyzed (Participants) | 2
changes in number of games played | -1.5 (.71)

6. Secondary Outcome: Changes in Gambling Frequency as Measured by Self Reported Frequency on 12 Different Types of Gambling
Description: as for outcome 1
Time Frame: Change from baseline to 12 months followup
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Non-Treatment: At the 12 month follow-up all people who completed the initial survey were again asked to complete the same measures. Only the baseline vs 12-month data is available.
Arm/Group | Online Treatment | Non-Treatment
Number analyzed (Participants) | 2 | 8
score on a scale | -4 (0) | -2.6 (3.4)

7. Secondary Outcome: Changes in Problem Gambling Severity Index (PGSI; Ferris & Wynne, 2001).
Description: as for outcome 2
Time Frame: Change from baseline to 12 months followup
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Treatment | Non-treatment
Number analyzed (Participants) | 2 | 8
score on a scale | -10 (2.83) | -8.3 (6.1)

8. Secondary Outcome: Changes in Kessler-6 (K6; Galea, et al., 2007).
Description: as for outcome 3
Time Frame: Change from baseline to 12 months followup
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Treatment | Non-treatment
Number analyzed (Participants) | 2 | 8
score on a scale | -3 (7) | -1.6 (5.4)

9. Secondary Outcome: Changes in Mindful Attention Awareness Scale (MAAS; Brown & Ryan, 2003).
Description: as for outcome 4
Time Frame: Change from baseline to 12 months followup
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Treatment | Non-treatment
Number analyzed (Participants) | 2 | 8
score on a scale | 1.1 (.05) | .32 (.84)

10. Secondary Outcome: Changes in Number of Games Played
Description: as for outcome 5
Time Frame: Change from baseline to 12 months followup
Measure: Mean (Standard Deviation); unit: changes in number of games played
Arm/Group | Online Treatment | Non-treatment
Number analyzed (Participants) | 2 | 8
changes in number of games played | -2.5 (.071) | -2.9 (2.7)

11. Other Pre Specified Outcome: Changes in Quality of lifeInventory (QLI) (Heun, et al., 2001)
Description: Higher levels of quality of life is expected as a result of the intervention. Each item was scored on a 6 point scale from "1, At no time" to "6, All of the time" for a total score ranging from 6 to 30. To assess the outcome we computed the difference score from pre-test to post-test which could range from 24 to -24 with positive numbers indicating improvement (higher quality of life).
Time Frame: Change from baseline to 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Treatment
Number analyzed (Participants) | 2
score on a scale | 2.0 (2.8)

12. Other Pre Specified Outcome: Changes in Quality of lifeInventory (QLI) (Heun, et al., 2001)
Description: as for outcome 11
Time Frame: Change from baseline to 12 months followup
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Treatment | Non-Treatment
Number analyzed (Participants) | 2 | 8
score on a scale | 2.0 (7.1) | 2.1 (3.8)

13. Other Pre Specified Outcome: Changes in Perceived Social Support (PSS) (Zimet et al., 1988)
Description: This scale measures perception of social support. Each item is measured on a 7 point scale from 1 to 7, for a total score of 12 to 84. Higher scores indicate higher levels of social support, so an increase in social support would be a positive change. For the evaluation we computer the differences from pre-test to post-test for a range from 72 to -72 with positive numbers indicate an improvement in perceived social support.
Time Frame: Change from baseline to 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Treatment
Number analyzed (Participants) | 2
score on a scale | -3.5 (7.8)

14. Other Pre Specified Outcome: Changes in Perceived Social Support (PSS) (Zimet et al., 1988)
Description: as for outcome 13
Time Frame: Change from baseline to 12 months followup
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Treatment | Non-treatment
Number analyzed (Participants) | 2 | 8
score on a scale | -3.5 (9.2) | 0.0 (14.1)

15. Other Pre Specified Outcome: Changes in The Random Events Knowledge Test (REKT)
Description: This scale measures the participants understanding of random events using a true or false format.. Each item is scored as correct or incorrect for a total score of 0 to 28. Higher scores mean they have a better understanding of random events and an increase in score would be a positive change. For the evaluation we computed the difference from pre-test to post-test for a range from 28 to -28 with positive number indicating improvement in the participants understanding of random chance.
Time Frame: Change from baseline to 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Treatment
Number analyzed (Participants) | 2
score on a scale | 3.5 (2.12)

16. Other Pre Specified Outcome: Changes in The Random Events Knowledge Test (REKT) Turner et al., (2006)
Description: as for outcome 15
Time Frame: Change from baseline to 12 months followup
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Treatment | Non-treatment
Number analyzed (Participants) | 2 | 8
score on a scale | 4 (1.41) | 0.5 (3.7)

17. Other Pre Specified Outcome: Changes in Visual Analog Scale of Cravings.
Description: The visual analog scale is based on similar measures used in drug research (e.g., Duncan, et al., 2001; Berger, et al., 1996). Each of 4 items is scored from 0 to 100, and the average is computed for a range from 0 to 100 with higher scores mean more cravings to gamble. A positive outcome would be lower scores at followup. For the evaluation we computed the difference between the post-test and pre-test for a range from 100 to -100, with negative numbers indicating an decrease in cravings.
Time Frame: Change from baseline to 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Treatment
Number analyzed (Participants) | 2
score on a scale | -9.63 (15.4)

18. Other Pre Specified Outcome: Changes in Visual Analog Scale of Cravings.
Description: as for outcome 17
Time Frame: Change from baseline to 12 months followup.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Treatment | Non-Treatment
Number analyzed (Participants) | 2 | 8
score on a scale | -25.5 (14.5) | -12.5 (31.9)

19. Other Pre Specified Outcome: Changes in Total Money Spent
Description: Self report measure of money spent gambling in past 6 months. Lower amounts spend would be a positive outcome.For the evaluation we compute the difference between spending at post-test from pre-test with negative numbers indicating an improvement (decrease in spending).
Time Frame: Change from baseline to 3 months
Measure: Mean (Standard Deviation); unit: change in dollars spent
Arm/Group | Online Treatment
Number analyzed (Participants) | 2
change in dollars spent | -3675 (2368)

20. Other Pre Specified Outcome: Changes in Total Money Spent
Description: as for outcome 19
Time Frame: Change from baseline to 12 months followup.
Measure: Mean (Standard Deviation); unit: change in dollars spent
Arm/Group | Online Treatment | Non-treatment
Number analyzed (Participants) | 2 | 8
change in dollars spent | -3750 (2474) | -3119 (4553)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Online Treatment
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

LIMITATIONS AND CAVEATS:
The main limitations of the current study is the small sample size and the absence of a randomly assigned control group. Due to the small sample size we examined the data in terms of two individual cases, rather than as a group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/85/NCT05084885/Prot_SAP_000.pdf